CLINICAL TRIAL: NCT01278992
Title: A Randomized Trial of Rhodiola Rosea for Mental and Physical Fatigue in Nurses
Brief Title: Rhodiola Rosea for Mental and Physical Fatigue
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Government of Alberta (Other Government)
Collaborators: University of Alberta (Other)
Responsible Party: Dr. Susan Lutz, Manager - Functional Foods and Natural Health Products, Government of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006C002P
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Fatigue
Keywords: fatigue; adaptogen; Rhodiola rosea
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Rhodiola rosea — 1 capsule = 182 mg Rhodiola rosea extract standardized to 2.8% total rosavins. Take 2 capsules at start of wakeful period each day. Participants will self-determine need for second dose, of 1 capsule, within 4 hours of the initial dose.
  Other Names: University of Alberta Lot Number 120910

SUMMARY:
The primary objective of this trial is to assess whether Rhodiola rosea improves fatigue when compared to placebo in nurses involved in shift work.

ELIGIBILITY:
Inclusion Criteria:

* Fourth year nursing students enrolled in NURS 495 (Nursing Practice)
* Participating in permanent overnight (between 11 pm and 7 am) or rotating shift work
* otherwise healthy
* consent to participate in the study

Exclusion Criteria:

* nurses aged 18 years or younger
* breastfeeding or pregnant women, as confirmed by a blood test
* female participants with child bearing potential not practicing a form of birth control throughout the trial
* presence of a primary medical condition associated with fatigue (e.g. cardiac, gastrointestinal, respiratory, renal, rheumatologic, or oncologic disease)
* presence of schizophrenia, bipolar disorder, dementia, eating disorders, insomnia or substance abuse
* presence of diabetes
* concurrent utilization of hypoglycaemic or agents for raising or lowering blood pressure
* known allergy or hypersensitivity to Rhodiola rosea or Sedum family extracts or pollen
* know allergy to microcrystalline cellulose or silicone dioxide
* concurrent utilization of stimulant drug such as methylphenidate (Ritalin), amphetamine (Dexedrine, Adderall), methamphetamine (Desoxyn) and pemoline (Cylert)
* concurrent utilization of other rhodiola or ginseng products (both fall in the same therapeutic category known as an "adaptogen")
* any significant medical condition
* any neurological or mental health condition
* taking medication that has central nervous system effects
* aged 55 years or older
* low blood pressure or history of significant dizziness

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 42 days
  A vitality subscale of the generic health-related quality of life instrument, RAND-36, will be employed to assess fatigue.
  A Visual Analogue Scale for Fatigue (VAS-F) will be concurrently administered to assess fatigue and compare to the RAND-36 fatigue assessment.

SECONDARY OUTCOMES:
Health-related quality of life | 42 days
  The health-related quality of life, RAND-36 will also assess physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social function, emotional well-being,and general health perceptions
Individualized Outcomes | 42 days
  Measure Yourself Medical Outcomes Profiles to measure change in items of importance to the participant, as identified by the participant.
Adaptive Capacity | 42 days
  Adaptive Capacity Index - 21 item questionnaire to measure a subject's ability to adapt to stressors
Adverse Event Monitoring | 42 days
  number of patients with any untoward medical occurance as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Vohra, MD FRCPC MSc, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Punja S, Shamseer L, Olson K, Vohra S. Rhodiola rosea for mental and physical fatigue in nursing students: a randomized controlled trial. PLoS One. 2014 Sep 30;9(9):e108416. doi: 10.1371/journal.pone.0108416. eCollection 2014. PMID 25268730